CLINICAL TRIAL: NCT05422677
Title: An Observational Study to Evaluate the Effectiveness and Safety of the Treatment of Tamsulosin in Korean Adult Males Diagnosed With Benign Prostatic Hyperplasia
Brief Title: An Observational Study of Tamsulosin in Patients With Benign Prostatic Hyperplasia
Status: Completed | Type: Observational
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: HM-TAM-OS-02
Record Dates: First submitted 2022-06-12; First posted 2022-06-16 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: BPH; Benign Prostatic Hyperplasia
Keywords: Tamsulosin; BPH; Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single arm, single group(No interventional): Observational
  Interventions: Drug: Hanmi Tams® Capsule

INTERVENTIONS:
Drug: Hanmi Tams® Capsule — Hanmi Tams®, Once daily administered per the locally approved product information

SUMMARY:
In this study, BPH patients visited the institutions during the study period and the effectiveness and safety of the treatment of Tamsulosin(Hanmi Tams® Capsule) in real-practice.

During the routine medical visit, according to the investigator's judgment, with diagnosis that the Tamsulosin prescription is appropriate, and after deciding to start treatment, patients with BPH who agreed to participate in the study were administered Tamsulosin.

As this study is a non-interventional observational study, all subjects received prescriptions according to the routine treatment procedure, and there were no visits or procedures required according to the observational study protocol.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, non-interventional, observational study of men administering Tamsulosin(Hanmi Tams® Capsule) to treat BPH.

Data will be collected from patients receiving routine treatment at hospitals in South Korea. Each subject visit the institution according to the protocol that designed the follow-up visits for six months to examine the effectiveness and safety of Tamsulosin.

This study will approved by the institutions' IRBs and is in compliance with clinical research ethics regulations.

ELIGIBILITY:
Inclusion Criteria:

* Male was diagnosed with Benign Prostatic Hyperplasia
* Those who first started taking Hanmi Tams®
* Those who voluntarily consented in writing to this study

Exclusion Criteria:

* Patients for whom use of Hanmi Tams® is prohibited

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Benign Prostatic Hyperplasia
Sampling Method: Non-Probability Sample
Enrollment: 4698 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
LUTS (Lower Tract Symptoms) improvement effect evaluated in patients with BPH symptoms after Tamsulosin treatment | 6 months
  To measure the level of LUTS (Lower Tract Symptoms), the IPSS was calculated.
  : The International Prostate Symptom Score (IPSS) is used to assess the severity of LUTS (Lower Tract Symptoms) and to monitor disease progression.
  The IPSS is calculated from 7 questions regarding incomplete emptying, frequency, intermittency, urgency, weak stream, and straining [rated as 0 (not at all) to 5 (almost always)], as well as how many times on average a participant has to get up to urinate at night (0=none to 5=5 times or more).
  The total score is classified as follows: 0 to 7 = mildly symptomatic; 8 to 19 = moderately symptomatic; and 20 to 35 = severely symptomatic.

CONTACTS AND LOCATIONS:
Overall Officials: Ji-yeon Hong, Study Director — Hanmi Pharmaceutical Company Limited
Locations (1):
- Hanmi Pharmaceutical Company Limited, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No